CLINICAL TRIAL: NCT04474821
Title: Acceptance and Completion Rate of Free HPV Vaccination Among Underserved Adult Patients (Age 18-45)
Brief Title: HPV Educational Intervention to Increase Acceptance and Completion of Free HPV Vaccination Among Underserved Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-010455; NCI-2020-04723 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 18-010455 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus Infection; Human Papillomavirus-Related Carcinoma
MeSH Terms: conditions — Papillomavirus Infections | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (HPV educational program) (Experimental): Patients receive educational materials on HPV and are asked of their willingness to proceed with the first HPV vaccination. Patients who express interest in receiving the HPV vaccination, then receive the first dose of the HPV vaccine and the next 2 doses approximately 2 months and 6 months following the initial vaccine.
  Interventions: Other: Educational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Educational Intervention — Receive educational materials on HPV
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase IV trial examines the impact of an education program on the human papilloma virus (HPV) and its effects on the acceptance and completion rates of a free HPV vaccination program in underserved adult patients. Participating in the HPV educational program may increase the HPV vaccination rates among low income uninsured adult patients and ultimately prevent HPV related cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the acceptability and completion rates of free HPV vaccination among the underserved adult patients at the Volunteer in Medicine Clinic (VIM) in Jacksonville, Florida.

II. Determine if an education program on HPV vaccination increases the acceptability of free HPV vaccination among the underserved adult patients at the Volunteer in Medicine Clinic (VIM) in Jacksonville, Florida.

III. Determine the baseline prevalence of HPV vaccination completion rates among VIM patients age 18-45.

IV. Determine if there are differences in acceptance and completion rates of HPV vaccination, among VIM patients of different sex, age (18-26 versus [vs] 27-45), ethnicity or race, following an education program on HPV as part of this protocol participation.

VI. Assessing possible barriers for vaccine series completion. VII. Determine if follow up intervention increases completion rate of free HPV vaccine series within 9 months.

OUTLINE:

Patients receive educational materials on HPV and are asked of their willingness to proceed with the first HPV vaccination. Patients who express interest in receiving the HPV vaccination, then receive the first dose of the HPV vaccine and the next 2 doses approximately 2 months and 6 months following the initial vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults patients seen at Volunteers in Medicine ages 18-45 years of age who read and understand English or Spanish

Exclusion Criteria:

* Children (under 18 years of age)
* Individuals who had previously received any dose of HPV vaccine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Acceptance and completion rates of free HPV vaccination | Up to 2 years

SECONDARY OUTCOMES:
Differences in acceptance and completion rates of HPV vaccination, among patients of different sex, ethnic or race | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Colon-Otero, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials